CLINICAL TRIAL: NCT06118671
Title: Application and Effectiveness Evaluation of Artificial Intelligence in Lifestyle Management of Diabetic Patients of Community
Brief Title: The Evaluation of Artificial Intelligence in Lifestyle Management of Diabetic Patients in Community
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Professor., Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BDT-CDR
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Diabetes
Keywords: lifestyle intervention; artificial intelligence
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): giving personalized lifestyle intervention suggestions through AI
  Interventions: Behavioral: personalized lifestyle intervention by AI
- Control group (No Intervention): giving routine lifestyle suggestions

INTERVENTIONS:
Behavioral: personalized lifestyle intervention by AI — The experimental group completed the basic information, diet structure, use of dietary supplements, living habits, and exercise according to the AI scale (AI scale can be entered through we-chat mini program search), and provided personalized lifestyle intervention plan according to the survey result.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn about the application and effectiveness evaluation of artificial intelligence (AI) in lifestyle management of diabetic patients in community.

DETAILED DESCRIPTION:
To determine the effectiveness of lifestyle intervention through AI on diabetic patients, whether it can improve blood sugar/ blood pressure/ body weight/ blood lipid control in people with type 1 or type 2 diabetes? Then find related risk factors. Participants will complete the basic information, diet structure, use of dietary supplements, living habits, and exercise according to the AI scale (AI scale can be entered through we-chat mini program search), and provided personalized lifestyle intervention plan according to the survey result, while the control group received routine lifestyle guidance. All included patients would fill in the patient's medication information according to the information content of the machine reading card, and follow up whether the medication is adjusted. The patient was included in the diabetes management we-chat group, followed up for 3 months /6 months according to the visit plan. The experimental group filled in the lifestyle assessment scale again, and personalized lifestyle intervention programs were provided according to the survey results, while the control group received routine follow-up and lifestyle guidance. Researchers will compare the two groups to see if the control of blood glucose, blood pressure, blood lipids and BMI of the experimental group after 6 months of AI-based lifestyle intervention was better than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Well informed of the procedures of this trial and informed consent is obtained
* 18-80 years old, gender is not limited
* Diagnosed diabetes (according to WHO1999 diagnostic criteria)
* Well compliance

Exclusion Criteria:

* Pregnant or lactating
* Poor blood glucose control (HbA1c>11%)
* A history of malignant tumor
* Abnormal liver or renal function [defined as alanine aminotransferase (ALT)>2.5 times higher than normal range, or eGFR<30 mL/min per 1.73 m2]
* Poor blood pressure control [systolic blood pressure (SBP)>180mmHg, or diastolic blood pressure (DBP)>110mmHg
* With severe heart disease, cardiac function worse than grade II, anemia (Hb<9.0g/d1)
* Blood routine test indicates that the white blood cell count (WBC) <3*109/L
* Body Mass Index (BMI)<18.5 or ≥35kg/m2
* Drug or alcohol abuse
* Accompanying mental disorder who can't collaborate
* Abnormal digestion and absorption function
* Other endocrine diseases
* Other chronic diseases needed long-term glucocorticoid treatment
* With severe infection, immune dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2023-11-07 (Estimated); Primary Completion 2024-11-07 (Estimated); Study Completion 2024-11-07 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1c | one year
  Change of HbA1c from baseline to endpoint (1 year follow-up)

SECONDARY OUTCOMES:
Change of systolic blood pressure | one year
  Change of systolic blood pressure from baseline to endpoint
Change of diastolic blood pressure | one year
  Reduction of diastolic blood pressure from baseline to endpoint
Change of LDL-c | one year
  Change of LDL-c from baseline to endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Hu, PhD, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- Jinbo Hu, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dobson R, Whittaker R, Jiang Y, Maddison R, Shepherd M, McNamara C, Cutfield R, Khanolkar M, Murphy R. Effectiveness of text message based, diabetes self management support programme (SMS4BG): two arm, parallel randomised controlled trial. BMJ. 2018 May 17;361:k1959. doi: 10.1136/bmj.k1959. PMID 29773539
- [Background] Wu Y, Min H, Li M, Shi Y, Ma A, Han Y, Gan Y, Guo X, Sun X. Effect of Artificial Intelligence-based Health Education Accurately Linking System (AI-HEALS) for Type 2 diabetes self-management: protocol for a mixed-methods study. BMC Public Health. 2023 Jul 11;23(1):1325. doi: 10.1186/s12889-023-16066-z. PMID 37434126
- [Background] Toi PL, Anothaisintawee T, Chaikledkaew U, Briones JR, Reutrakul S, Thakkinstian A. Preventive Role of Diet Interventions and Dietary Factors in Type 2 Diabetes Mellitus: An Umbrella Review. Nutrients. 2020 Sep 6;12(9):2722. doi: 10.3390/nu12092722. PMID 32899917
- [Background] Viguiliouk E, Kendall CW, Kahleova H, Rahelic D, Salas-Salvado J, Choo VL, Mejia SB, Stewart SE, Leiter LA, Jenkins DJ, Sievenpiper JL. Effect of vegetarian dietary patterns on cardiometabolic risk factors in diabetes: A systematic review and meta-analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1133-1145. doi: 10.1016/j.clnu.2018.05.032. Epub 2018 Jun 13. PMID 29960809
- [Background] Nundy S, Dick JJ, Chou CH, Nocon RS, Chin MH, Peek ME. Mobile phone diabetes project led to improved glycemic control and net savings for Chicago plan participants. Health Aff (Millwood). 2014 Feb;33(2):265-72. doi: 10.1377/hlthaff.2013.0589. PMID 24493770
- [Background] Arambepola C, Ricci-Cabello I, Manikavasagam P, Roberts N, French DP, Farmer A. The Impact of Automated Brief Messages Promoting Lifestyle Changes Delivered Via Mobile Devices to People with Type 2 Diabetes: A Systematic Literature Review and Meta-Analysis of Controlled Trials. J Med Internet Res. 2016 Apr 19;18(4):e86. doi: 10.2196/jmir.5425. PMID 27095386
- [Background] Sarkar U, Karter AJ, Liu JY, Adler NE, Nguyen R, Lopez A, Schillinger D. The literacy divide: health literacy and the use of an internet-based patient portal in an integrated health system-results from the diabetes study of northern California (DISTANCE). J Health Commun. 2010;15 Suppl 2(Suppl 2):183-96. doi: 10.1080/10810730.2010.499988. PMID 20845203
- [Background] Chiavaroli L, Lee D, Ahmed A, Cheung A, Khan TA, Blanco S, Mejia, Mirrahimi A, Jenkins DJA, Livesey G, Wolever TMS, Rahelic D, Kahleova H, Salas-Salvado J, Kendall CWC, Sievenpiper JL. Effect of low glycaemic index or load dietary patterns on glycaemic control and cardiometabolic risk factors in diabetes: systematic review and meta-analysis of randomised controlled trials. BMJ. 2021 Aug 4;374:n1651. doi: 10.1136/bmj.n1651. PMID 34348965
- [Background] Wagner EH, Sandhu N, Newton KM, McCulloch DK, Ramsey SD, Grothaus LC. Effect of improved glycemic control on health care costs and utilization. JAMA. 2001 Jan 10;285(2):182-9. doi: 10.1001/jama.285.2.182. PMID 11176811